CLINICAL TRIAL: NCT01341405
Title: A Double-blind, Randomized, Multicenter, Noninferiority, Phase II Repeat Dose Study of CG100649 Versus Celecoxib in Osteoarthritis Patients
Brief Title: Study of CG100649 Versus Celecoxib in Osteoarthritis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CrystalGenomics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CG100649-2-02
Record Dates: First submitted 2011-04-22; First posted 2011-04-25 (Estimated); Results first posted 2023-02-09 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2022-05

CONDITIONS: Osteoarthritis
Keywords: COX-1; COX-2; carbonic anhydrase; anti-inflammatory; Cyclooxygenase Inhibitors; Polmacoxib
MeSH Terms: conditions — Osteoarthritis | interventions — CG100649; Celecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CG100649 2 mg (Experimental): capsule, once daily for 28 days
  Interventions: Drug: CG100649
- CG100649 4 mg (Experimental): capsule, once daily for 28 days
  Interventions: Drug: CG100649
- celecoxib 200 mg (Active Comparator): capsule, once daily for 28 days
  Interventions: Drug: Celecoxib

INTERVENTIONS:
Drug: CG100649 — once daily for 28 days
  Other Names: CG100649 2mg; CG100649 4mg
  Arms: CG100649 2 mg; CG100649 4 mg
Drug: Celecoxib — capsule, celecoxib 200 mg, once daily for 28 days
  Other Names: Celebrex
  Arms: celecoxib 200 mg

SUMMARY:
This is a double-blind, randomized, multicenter, phase 2b, noninferiority comparison of two active dose levels of CG100649 vs. a standard anti-arthritic dose of celecoxib (Celebrex).

DETAILED DESCRIPTION:
This is a double-blind, randomized, multicenter, noninferiority, phase 2 study. Subjects will discontinue current medications (NSAID or COX-2 inhibitor) 5-14 days prior to randomization. Paracetamol (acetaminophen; ≤2 gm/day) may be used for breakthrough pain. Other NSAIDs, COX-2 inhibitors, opioids, and corticosteroids may not be used at any time during this study. Only subjects recording average WOMAC pain score of 4 to 8 on a 0-10 numerical rating scale during the washout period and meeting all other inclusion criteria will be randomized into the study.

Male and female adults, ages 20 and older, with a history of osteoarthritis (OA) of the knee or hip diagnosed by radiograph obtained within the past 20 years and with pain at least 3 months from OA can participate in this study. OA must be confirmed by radiographs and diagnosed according to American College of Rheumatology (ACR) guidelines. Subjects must qualify as ACR global functional status I, II, or III (excluding IV) and Kellgren-Lawrence grade 1, 2 or 3 (excluding grade 4).

Subjects meeting screening criteria will be randomized to receive 28 days dosing of an active dose of CG100649 or comparator (celecoxib).

Antiarthritic efficacy will be evaluated by changes in the Western Ontario and McMaster Universities (WOMAC) OA index completed on Day 1 (Baseline) and on Days 14, 28 and 42. The WOMAC pain subscale will be evaluated at screening and on Days 1, 7, 14, 21, 28, 35 and 42.

All doses will be administered orally once daily in the morning. There are 3 planned treatment arms (2 with active compound + one comparator (celecoxib) group) with n=44 per treatment arm. Total number of subjects will be 132.

Treatment A: CG100649: 2 mg/day (Days 1-28); Treatment B: CG100649: 4 mg/day (Days 1-28); Treatment C: celecoxib: 200 mg/day (Days 1-28); Active and comparator medications will have identical appearance.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 20 years old and more, able and willing to provide written informed consent to participate in the study
2. Confirmed osteoarthritis (OA) of the knee or hip by radiograph obtained within the past 20 years and diagnosed according to American College of Rheumatology (ACR) guidelines.
3. Subject must have pain at least 3 month duration from osteoarthritis (OA)
4. Normal blood pressure (BP) [systolic BP 90-140 mmHg, diastolic BP 50-90 mmHg] and heart rate (HR) [resting 45-90 beats per minute (bpm)]
5. Subjects with hypertension should have stably taken ACE inhibitor, angiotensin II receptor (type AT1) antagonist, beta-blocker and/or diuretics at least 3 months at the time of screening in order to keep normal blood pressure. Subjects should not change or stop hypertension drug during the study.
6. Clinical Chemistry must be within 2x normal limits
7. Urinalysis must be within normal range.
8. Prior to randomization on Day 1, the mean WOMAC pain score in the index joint must be between 4 and 8 on a 0-10 numerical rating scale.
9. Subjects and their sexual partners must agree to use double barrier contraception during the study period and for 3 months afterwards or provide proof of surgical sterility or post-menopause more than 1 year.
10. Subject must be able to read and understand and follow the study instructions.

Exclusion Criteria:

1. Use of any analgesics except the study medication or paracetamol (acetaminophen) at any time during this study;
2. Use of corticosteroids or intra-articular viscosupplementation within 3 months of screening;
3. Use of antidepressants or anticonvulsants within 2 months of screening;
4. Cognitive or psychiatric disorders, or daytime use of medications (alcohol, benzodiazepines, barbiturates, muscle relaxants) that could diminish compliance with study procedures;
5. Use of anticoagulants (aspirin, warfarin, heparin) within 2 weeks of screening;
6. Use of any medications that will affect pain perception (e.g. tranquilizers, hypnotics);
7. Hypersensitivity to non-steroidal anti-inflammatory drugs (NSAIDs), cyclooxygenase (COX)-2 inhibitors, or carbonic anhydrase inhibitors;
8. Use of oriental medicine (herbal medicine) or glucosamine within 14 days of dose administration
9. History of drug or alcohol abuse within one year prior to screening;
10. Known allergy or hypersensitivity to sulfa drugs;
11. History of congestive heart failure, ischemic heart disease, peripheral arterial disease, cerebrovascular disease or subjects who have one of these diseases;
12. Use of chemotherapy agents or history of cancer, other than non-metastatic skin cancer that has been completely excised, within five (5) years prior to the screening visit;
13. Subjects with gout, pseudogout, inflammatory arthritis, Paget's disease, chronic pain syndrome, fibromyalgia, or another major joint disease;
14. Subjects requiring knee or hip arthroplasty within 2 months of screening or anticipating any need for a surgical procedure on the index joint during the study;
15. Subjects who have had surgery on the affected joint within 6 months of screening and subjects with a prosthesis at the index joint;
16. History of seizure disorder;
17. Subjects with serious psychosocial co-morbidities;
18. Subjects with gastrointestinal, renal, hepatic, or coagulant disorder within 6 months of screening;
19. Esophageal or duodenal ulcer within 6 months of screening;
20. History of nasal polyps, bronchospasm, and urticaria;
21. Pregnant or breast-feeding;
22. Subject with genetic problem of galactose intolerance, Lapp lactose deficiency or glucose-galactose malabsorption (because celecoxib contains lactose)

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2011-04; Primary Completion 2011-12 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sangsook Cho, Ph.D., Study Director — CrystalGenomics, Inc.
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from Apr 2011 to Dec 2011 in 5 sites in Korea.
Groups:
- CG100649 2 mg; CG100649 4 mg; Celecoxib 200 mg: once daily for 28 days
Period: Overall Study
Arm/Group | CG100649 2 mg | CG100649 4 mg | Celecoxib 200 mg
Started | 40 | 42 | 43
Completed | 37 | 39 | 41
Not Completed | 3 | 3 | 2
Not completed — Adverse Event | 0 | 1 | 1
Not completed — Withdrawal by Subject | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CG100649 2 mg | CG100649 4 mg | Celecoxib 200 mg | Total
Number analyzed (Participants) | 40 | 42 | 43 | 125
Age, Continuous [Mean (Standard Deviation); unit: years]
  Age | 62.1 (8.24) | 59 (7.48) | 61 (7.51) | 60.7 (7.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 37 | 39 | 112
  Male | 4 | 5 | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change of the WOMAC Pain Subscale at Day 28 From Baseline
Description: Changes in the WOMAC Pain Score from Baseline The primary endpoint of this study was the change in the sum of the WOMAC Pain subscale at Day 28 vs. Baseline (Day 1) using the ITT population). Pain scores were evaluated using the WOMAC Pain subscale, which provided an evaluation of pain during the past 48 hours using a 0-10 numerical rating scale for each of 5 questions (minimum total: 0 point, maximum total: 50 points). A higher WOMAC Pain score represented worse symptom severity.
Time Frame: Baseline, Day 28
Population: intent-to-treat population (BOCF)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- CG100649 2mg; CG100649 4mg; Celecoxib 200 mg: once daily for 28 days
Arm/Group | CG100649 2mg | CG100649 4mg | Celecoxib 200 mg
Number analyzed (Participants) | 40 | 42 | 43
units on a scale | -14.33 [-16.70 to -11.97] | -12.47 [-14.89 to -10.05] | -13.24 [-15.73 to -10.76]

2. Secondary Outcome: Change of the Sum of WOMAC OA Index at Day 28 From Baseline
Description: The numerical rating scale version of the Western Ontario and McMaster Universities (WOMAC) OA index will be used-i.e., with the patient assessing each question by a 11-point (0-10) numerical rating scale, and the total index score being represented by the sum of the 24 component item scores. A higher WOMAC score represents worse symptom severity, with 240 being the worst possible total score (minimum total: 0 point, maximum total: 240 points).
Time Frame: Baseline, Day 28
Population: intent-to-treat population (BOCF)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CG100649 2mg | CG100649 4mg | Celecoxib 200 mg
Number analyzed (Participants) | 40 | 42 | 43
units on a scale | -49.94 [-60.65 to -39.23] | -41.61 [-52.81 to -30.40] | -43.80 [-53.52 to -34.09]

3. Secondary Outcome: Change of WOMAC-Stiffness Subscale at Day 28 From Baseline
Description: Version 3.1 of the WOMAC knee and hip osteoarthritis index translated in Korean language was used to evaluate the stiffness of the index joint. Two questions were to evaluate "Stiffness" of the index joint. A higher WOMAC-Stiffness score represents worse symptom severity, with 20 being the worst possible total score (minimum total: 0 point, maximum total: 20 points).
Time Frame: Baseline, Day 28
Population: intent-to-treat population (BOCF)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CG100649 2mg | CG100649 4mg | Celecoxib 200 mg
Number analyzed (Participants) | 40 | 42 | 43
units on a scale | -3.17 [-4.33 to -2.00] | -2.87 [-4.02 to -1.71] | -2.32 [-3.29 to -1.34]

4. Secondary Outcome: Change of WOMAC-Physical Function Subscale at Day 28 From Baseline
Description: Version 3.1 of the WOMAC knee and hip osteoarthritis index translated in Korean language was used. The total 17 questions to evaluate "Physical Function." A higher score of WOMAC-Physical function subscale represents worse symptom severity, with 170 being the worst possible total score (minimum total: 0 point, maximum total: 170 points).
Time Frame: Baseline, Day 28
Population: intent-to-treat population (BOCF)
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | CG100649 2mg | CG100649 4mg | Celecoxib 200 mg
Number analyzed (Participants) | 40 | 42 | 43
units on a scale | -32.44 [-40.44 to -24.45] | -26.26 [-34.77 to -17.75] | -28.24 [-35.47 to -21.02]

ADVERSE EVENTS:
Time Frame: from ICF to treatment completion
Groups:
- CG100649 4mg,: once daily for 28 days
- Celecoxib 200mg: once daily for 28 dyas
Arm/Group | CG100649 2mg | CG100649 4mg, | Celecoxib 200mg
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/42 | 0/43
Other Adverse Events (participants affected / at risk) | 13/40 | 22/42 | 10/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CG100649 2mg (N=40) | CG100649 4mg, (N=42) | Celecoxib 200mg (N=43)
Abdominal Pain Upper (Gastrointestinal disorders) | 3 (3) | 6 (6) | 3 (3)
Dyspepsia (Gastrointestinal disorders) | 4 (4) | 9 (9) | 3 (3)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 3 (3)
chest discomfort (General disorders) | 0 (0) | 3 (3) | 0 (0)
face edema (General disorders) | 1 (1) | 3 (3) | 0 (0)
Oropharyngeal pain (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication requires prior expressed written consent of Sponsor.